CLINICAL TRIAL: NCT01413672
Title: Peristomal Skin Irritation: A Preliminary Evaluation of CASTLE Barrier North American Prototype
Brief Title: Preliminary Evaluation of CASTLE Barrier North American Prototype
Status: Completed | Type: Observational
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 5075-O
Record Dates: First submitted 2011-08-06; First posted 2011-08-10 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Peristomal Skin Complication
Keywords: ostomy; colostomy; ileostomy; barrier; irritation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- person with ostomy: Community dwelling subject with either colostomy or ileostomy and at least 3 months post-surgery.
  Interventions: Device: Use of CASTLE barrier

INTERVENTIONS:
Device: Use of CASTLE barrier — Test barrier to be used in place of normal barrier. Otherwise normal routine is followed

SUMMARY:
The purpose of this study is to determine if an ostomy barrier that promotes a healthy skin environment will result in reduced peristomal skin irritation.

ELIGIBILITY:
Inclusion Criteria:

at least 18 years of age has colostomy or ileostomy current user of two-piece, flat, tape bordered barrier mild to moderate skin peristomal skin irritation community dwelling and cares for stoma independently at least 3 months post-operative provides informed consent

Exclusion Criteria:

presence of fistula on or near stoma prior participation in stoma care study within past 30 days pregnant or lactating (interview only) uses convex product, paste and/or rings known allergy to test barrier composition existing medical condition or therapy that might affect ability to participate or interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects currently known to investigators
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Peristomal skin irritation | 30 days

SECONDARY OUTCOMES:
Security | 30 days
  wear time, lifting of barrier from skin, leakage

CONTACTS AND LOCATIONS:
Overall Officials: Richard Murahata, Ph.D., Study Director — Hollister Incorporated
Locations (5):
- United States (4):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - ET Nursing Services, Jacksonville, Florida
  - St. Louis Medical, Fenton, Missouri
  - Restored Images, Kansas City, Missouri
- Ostomy Care & Supply Centre, New Westminster, British Columbia, Canada